CLINICAL TRIAL: NCT00107653
Title: A Prospective, Multicenter, Open-label, Comparative, Efficacy Study of Pegasys® Plus Copegus® in Treatment-naïve Latino Patients With Chronic Hepatitis C-genotype 1, as Compared to Treatment-naïve Non- Latino Caucasian Patients With Chronic Hepatitis C-genotype 1
Brief Title: Latino Study - A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) and COPEGUS (Ribavirin) in Treatment-Naive Patients With Chronic Hepatitis C-Genotype 1.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18179
Record Dates: First submitted 2005-04-06; First posted 2005-04-07 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (2):
- Latino (Experimental): Participants received peginterferon alfa-2a 180 microgram (mcg)/0.5 mL by subcutaneous injection once a week in combination with ribavirin 1000 or 1200 mg per day, which was taken orally in split doses for 48 weeks. Participants with <75 kg (165 lbs) of body weight received 1000 mg/day (400 mg in the morning and 600 mg in the evening). Participants with >=75 kg (165 lbs) of body weight received 1200 mg/day (600 mg in the morning and 600 mg in the evening).
  Interventions: Drug: Ribavirin; Drug: Peginterferon alfa-2a
- Non-Latino White (Experimental): Participants received peginterferon alfa-2a 180 mcg/0.5 mL by subcutaneous injection once a week in combination with ribavirin 1000 or 1200 mg per day which was taken orally in split doses. Participants with <75 kg (165 lbs) of body weight received 1000 mg/day. Participants with >=75 kg (165 lbs) of body weight received 1200 mg/day for 48 weeks.
  Interventions: Drug: Ribavirin; Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Ribavirin — 1000-1200mg po daily for 48 weeks
  Arms: Latino
Drug: Peginterferon alfa-2a — 180 micrograms sc/week for 48 weeks
  Arms: Latino
Drug: Ribavirin — 1000-1200mg po daily for 48 weeks
  Arms: Non-Latino White
Drug: Peginterferon alfa-2a — 180 micrograms sc/week for 48 weeks
  Arms: Non-Latino White

SUMMARY:
This single arm study will evaluate the efficacy and safety of PEGASYS (180 micrograms sc weekly) plus ribavirin (1000-1200mg po daily) in treatment-naive Latino patients versus non-Latino Caucasian patients with chronic hepatitis C- genotype 1. The anticipated time on study treatment is 3-12 months and the target sample size is 500+ patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-65 years of age
* chronic hepatitis C , genotype 1
* serologic evidence of CHC infection by an antibody test
* chronic liver disease, consistent with CHC infection on a liver biopsy obtained within the past 18 months
* compensated liver disease
* use of 2 forms of contraception during the study in both men and women

Exclusion Criteria:

* previous interferon or ribavirin therapy
* systemic antiviral therapy less than 24 weeks before first dose of study drug or expected need for this treatment any time during the study
* medical condition associated with chronic liver disease (eg, hemochromatosis, autoimmune hepatitis, alcoholic liver disease, toxin exposure)
* decompensated liver disease
* women who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- United States (49):
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Fountain Valley, California
  - Fresno, California
  - Lancaster, California
  - Los Angeles, California
  - Palo Alto, California
  - Redlands, California
  - Sacramento, California
  - San Bernardino, California
  - San Diego, California
  - San Francisco, California
  - San Luis Obispo, California
  - Ventura, California
  - Pueblo, Colorado
  - Boca Raton, Florida
  - Bradenton, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - Plantation, Florida
  - Austell, Georgia
  - Chicago, Illinois
  - Gurnee, Illinois
  - Indianapolis, Indiana
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Framingham, Massachusetts
  - Worcester, Massachusetts
  - St Louis, Missouri
  - Vineland, New Jersey
  - Bayside, New York
  - New York, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Fayetteville, North Carolina
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Sam Houston, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Seattle, Washington
  - Tacoma, Washington
- Puerto Rico (2):
  - Ponce
  - Santurce

REFERENCES:
- [Derived] Rodriguez-Torres M, Jeffers LJ, Sheikh MY, Rossaro L, Ankoma-Sey V, Hamzeh FM, Martin P; Latino Study Group. Peginterferon alfa-2a and ribavirin in Latino and non-Latino whites with hepatitis C. N Engl J Med. 2009 Jan 15;360(3):257-67. doi: 10.1056/NEJMoa0805062. PMID 19144941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 569 participants were recruited at 52 centers in the United States in the study conducted from 26 October 2004 and 07 September 2007.
Pre-assignment Details: Out of 1038 screened participants, 569 were enrolled and 469 were screen failures because of eligibility criteria was not met. Of the 569 enrolled participants, 269 participants were assigned to Latino and 300 participants were assigned to non-Latino White group.
Groups:
- Latino: Eligible participants received peginterferon alfa-2a 180 microgram (mcg)/0.5 mL by subcutaneous injection once a week in combination with ribavirin 1000 or 1200 mg per day, which was taken orally in split doses for 48 weeks. Participants with <75 kg (165 lbs) of body weight received 1000 mg/day (400 mg in the morning and 600 mg in the evening). Participants with >=75 kg (165 lbs) of body weight received 1200 mg/day (600 mg in the morning and 600 mg in the evening).
- Non-Latino White: Eligible participants received peginterferon alfa-2a 180 mcg/0.5 mL by subcutaneous injection once a week in combination with ribavirin 1000 or 1200 mg per day which was taken orally in split doses. Participants with <75 kg (165 lbs) of body weight received 1000 mg/day. Participants with >=75 kg (165 lbs) of body weight received 1200 mg/day for 48 weeks.
Period: Overall Study
Arm/Group | Latino | Non-Latino White
Started | 269 | 300
Completed | 190 | 224
Not Completed | 79 | 76
Not completed — Adverse Event | 24 | 43
Not completed — Insufficient Therapeutic Response | 25 | 11
Not completed — Violation of Selection Criteria at Entry | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 12 | 13
Not completed — Lost to Follow-up | 13 | 5
Not completed — Administrative Reasons | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Latino | Non-Latino White | Total
Number analyzed (Participants) | 269 | 300 | 569
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (8.79) | 48.1 (8.34) | 46.9 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 108 | 194
  Male | 183 | 192 | 375

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at Week 72
Description: Sustained Virologic Response (SVR) is defined as percentage of participants with an undetectable hepatitis C virus-RNA (HCV-RNA) measurement (<28 International Unit (IU)/millilitre (mL)) assessed 24 weeks post-treatment (week 72) which was assessed by Roche High Pure System/COBAS TaqMan HCV Test.
Time Frame: At Week 72
Population: Intent-to-Treat (ITT) Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus).
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 300
Percentage of participants | 33.5 | 49.3
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; SVR for Latino Versus (VS) Non-Latino White; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial. — P-values are calculated based on the difference in proportion between Latino and Non-Latino White group; SVR for Study Group Difference = -0.16, 95% CI 2-sided [-0.24 to -0.08], Standard Error of Mean 0.041 — The estimated value is the difference in proportion of participants (Latino minus Non-Latino White) with SVR. The 95% Confidence Interval is based on normal approximation to the binomial

2. Secondary Outcome: Percentage of Participants Achieving Virologic Response
Description: Percentage of participants achieving a virologic response defined as an undetectable HCV-RNA measurement (HCV-RNA <28 IU/mL by Roche High Pure System/COBAS TaqMan HCV Test)
Time Frame: At Weeks 4, 12, 24, 48, 60, and 72
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus).
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 300
Percentage of participants
  At Week 4 | 13.8 | 20.0
  At Week 12 | 48.0 | 63.0
  At Week 24 | 59.5 | 73.3
  At Week 48 | 56.1 | 72.7
  At Week 60 | 33.1 | 50.0
  At Week 72 | 33.5 | 49.3
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 4; Test type: Superiority or Other; p = 0.0454, Normal approximation to the binomial; Study Group Difference = -0.06, 95% CI 2-sided [-0.12 to -0.00], Standard Error of Mean 0.031 — The estimated value is the difference in proportion of participants (Latino minus Non-Latino White) with virologic response. The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 12; Test type: Superiority or Other; p = 0.0003, Normal approximation to the binomial; Study Group Difference = -0.15, 95% CI 2-sided [-0.23 to -0.07], Standard Error of Mean 0.041 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 24; Test type: Superiority or Other; p = 0.0004, Normal approximation to the binomial; Study Group Difference = -0.14, 95% CI 2-sided [-0.22 to -0.06], Standard Error of Mean 0.039 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 48; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = -0.17, 95% CI 2-sided [-0.24 to -0.09], Standard Error of Mean 0.040 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 60; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = -0.17, 95% CI 2-sided [-0.25 to -0.09], Standard Error of Mean 0.041 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 72; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = -0.16, 95% CI 2-sided [-0.24 to -0.08], Standard Error of Mean 0.041 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With Early Virologic Response at Week 4
Description: Percentage of participants with an early virologic response defined as an HCVRNA >=1 log10 drop from baseline or undetectable HCV-RNA measurement at Week 4 (lower limit of detection 28 IU/mL).
Time Frame: At Week 4
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus).
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 300
Percentage of participants | 71.0 | 78.7
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 4; Test type: Superiority or Other; p = 0.0353, Normal approximation to the binomial; Study Group Difference = -0.08, 95% CI 2-sided [-0.15 to -0.01], Standard Error of Mean 0.036 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With Early Virologic Response at Week 12
Description: Percentage of participants with an early virologic response defined as an HCV-RNA >=2 log10 drop from baseline or undetectable HCV-RNA measurement at Week 12 (lower limit of detection 28 IU/mL).
Time Frame: At Week 12
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus).
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 300
Percentage of participants | 75.5 | 86.0
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; Virologic Response for Latino VS Non-Latino White at Week 12; Test type: Superiority or Other; p = 0.0014, Normal approximation to the binomial; Study Group Difference = -0.11, 95% CI 2-sided [-0.17 to -0.04], Standard Error of Mean 0.033 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in HCV-RNA Log10 Titers Over the Period Of Time
Description: The table below shows HCV-RNA log10 titers change from baseline values by study week and by study group. Analysis was performed for participants with a baseline and at least 1 post-baseline HCV-RNA assessment. HCV-RNA quantitation was performed using Roche High Pure System/COBAS® TaqMan® HCV Monitor Test. HCV-RNA measurement lower limit of detection was 28 IU/mL.
Time Frame: From Baseline (Week 0) to Weeks 4, 12, 24, 48, 60 and 72
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus). 'n'=number of evaluable participants available at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Log10 IU/mL
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 262 | 280
Log10 IU/mL
  At Week 4 (n=262, 280) | -2.3 (0.10) | -2.9 (0.09)
  At Week 12 (n=251,279) | -3.9 (0.10) | -4.5 (0.09)
  At Week 24 (n=235, 264) | -4.2 (0.11) | -4.8 (0.10)
  At Week 48 (n=207, 246) | -4.1 (0.11) | -4.8 (0.10)
  At Week 60 (n=181, 217) | -2.7 (0.17) | -3.7 (0.15)
  At Week 72 (n=174, 212) | -2.7 (0.17) | -3.6 (0.16)

6. Secondary Outcome: Percentage of Participants With Biochemical Response
Description: Biochemical response was defined as normal serum alanine transaminase (ALT) measurement. For ALT measurement the normal range is 5-37 IU/L.
Time Frame: At Weeks 4, 12, 24, 48, 60 and 72
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus).
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 300
Percentage of participants
  At Week 4 | 42.8 | 57.0
  At Week 12 | 56.1 | 72.0
  At Week 24 | 53.2 | 68.0
  At Week 48 | 45.7 | 59.7
  At Week 60 | 35.3 | 53.7
  At Week 72 | 37.5 | 56.7
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; Normal Serum ALT level for Latino VS Non-Latino White at Week 4; Test type: Superiority or Other; p = 0.0006, Normal approximation to the binomial; Study Group Difference = -0.14, 95% CI 2-sided [-0.22 to -0.06], Standard Error of Mean 0.042 — The estimated value is the difference in proportion of participants (Latino minus Non-Latino White) with biochemical response. The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Latino vs Non-Latino White; Normal Serum ALT level for Latino VS Non-Latino White at Week 12; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = -0.16, 95% CI 2-sided [-0.24 to -0.08], Standard Error of Mean 0.040 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Latino vs Non-Latino White; Normal Serum ALT level for Latino VS Non-Latino White at Week 24; Test type: Superiority or Other; p = 0.0003, Normal approximation to the binomial; Study Group Difference = -0.15, 95% CI 2-sided [-0.23 to -0.07], Standard Error of Mean 0.041 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Latino vs Non-Latino White; Normal Serum ALT level for Latino VS Non-Latino White at Week 48; Test type: Superiority or Other; p = 0.0008, Normal approximation to the binomial; Study Group Difference = -0.14, 95% CI 2-sided [-0.22 to -0.06], Standard Error of Mean 0.042 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Latino vs Non-Latino White; Normal Serum ALT level for Latino VS Non-Latino White at Week 60; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = -0.18, 95% CI 2-sided [-0.26 to -0.10], Standard Error of Mean 0.041 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Latino vs Non-Latino White; Normal Serum ALT level for Latino VS Non-Latino White at Week 72; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = -0.19, 95% CI 2-sided [-0.27 to -0.11], Standard Error of Mean 0.041 — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Percentage of Participants With ISHAK Histological Activity Index Response
Description: ISHAK Histological Activity Index (HAI) activity response is defined as a decrease from baseline of at least 2 points (≥2 points drop from baseline) in the ISHAK modified HAI (necroinflammatory) score at week 72. ISHAK modified HAI activity (necroinflammatory) score is a total score of periportal ± bridging (P/B) necrosis + confluent necrosis + focal necrosis + portal inflammation (maximum score for each participant = 18). Where P/B necrosis grading as 0 = absent; 1 = mild; 2 = mild/moderate; 3 = moderate; 4 = severe; Confluent necrosis grading as 0 = absent; 1 = focal; 2 = zone 3 some areas; 3 = zone 3 most areas; 4 = zone 3 occasional portal; 5 = zone 3 multiple; 6 = panacinar necrosis and Focal necrosis grading as 0: absent; 1: < = 1 focus; 2: 2 to 4 foci; 3: 5 to 10 foci; 4: > 10 foci; Portal Inflammation grading: 0 = none; 1 = mild; 2 = moderate; 3 = moderate/marked; 4 = marked/all portal.
Time Frame: At Week 72
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus). Analysis was performed for ITT participants with paired biopsy.
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Percentage of participants | 47.1 | 58.7
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; ISHAK HAI Response For Latino VS Non-Latino White; Test type: Superiority or Other; p = 0.0285, Normal approximation to the binomial; Study Group Difference = -0.12, 95% CI 2-sided [-0.2 to -0.0], Standard Error of Mean 0.05 — The estimated value is the difference in proportion of participants (Latino minus Non-Latino White) with ISHAK HAI response. The 95% Confidence Interval is based on normal approximation to the binomial

8. Secondary Outcome: Mean Change From Baseline in ISHAK HAI Activity (Necroinflammatory) at Week 72
Description: ISHAK modified HAI activity (necroinflammatory) score is a total score of P/B necrosis + confluent necrosis + focal necrosis + portal inflammation (maximum score for each Participant = 18). Where P/B necrosis grading as 0 = absent; 1 = mild; 2 = mild/moderate; 3 = moderate; 4 = severe; Confluent necrosis as 0 = absent; 1 = focal; 2 = zone 3 some areas; 3 = zone 3 most areas; 4 = zone 3 occasional portal; 5= zone 3 multiple; 6= panacinar necrosis and Focal necrosis as 0: absent; 1: <= 1 focus; 2: 2 to 4 foci; 3: 5 to 10 foci; 4: > 10 foci; Portal Inflammation: 0 = none; 1 = mild; 2 = moderate; 3 = moderate/marked; 4 = marked/all portal. The difference between study groups in change from baseline in ISHAK modified HAI activity score at week 72 was tested using an analysis of covariance (ANCOVA) model with ethnicity and baseline ISHAK HAI score as the fixed effects.
Time Frame: From Baseline (Week 0) to Week 72
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Score on a scale | -1.4 (0.17) | -2.1 (0.17)
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; ISHAK HAI activity For Latino VS Non-Latino White; Test type: Superiority or Other; p < 0.0001, Normal approximation to the binomial; Study Group Difference = 0.9, 95% CI 2-sided [0.5 to 1.3], Standard Error of Mean 0.20 — The estimated value is the difference in change from baseline of ISHAK HAI activity (necroinflammatory) scores between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial

9. Secondary Outcome: Mean Change From Baseline in Fibrosis Score Based on ISHAK at Week 72
Description: ISHAK Histological Activity Index (HAI) activity response is defined as a decrease from baseline of at least 2 points (≥2 points drop from baseline) score at week 72. Baseline prognostic factors in the original model include ethnicity, sex, age, baseline ALT quotient, baseline HCV-RNA level, and ISHAK fibrosis and activity scores at baseline. ISHAK modified HAI fibrosis scale by fibrosis grading category as F0= no fibrosis; F1= some portal areas; F2= most portal areas; F3= bridging fibrosis; F4= bridging and portal to central; F5 = marked bridging; F6 = Cirrhosis; where '0' being the best and '6' being the worst. Decrease in score from baseline indicates improvement. The difference between study groups in change from baseline in ISHAK modified HAI activity score at week 72 was analysed.
Time Frame: From Baseline (Week 0) to Week 72
Population: ITT Population included all participants who were enrolled and took at least 1 dose of study drug (Pegasys or Copegus). Analysis was performed for ITT participants with paired biopsy. 'n'=number of evaluable participants available at specified time point.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Score on a scale
  F5-F6 (n=21,11) | -1.05 (0.42) | -2.64 (0.82)
  F0-F4 (n=136,190) | -1.49 (0.19) | -2.04 (0.18)

10. Secondary Outcome: Percentage of Participants With Improved, Stable and Worsened ISHAK Fibrosis Score
Description: Overall ISHAK Fibrosis Score is defined as Improved: >= 1 category decrease in fibrosis scale; Stable: no change in fibrosis scale; Worsened: >1 category increase in fibrosis scale.
Time Frame: At Week 72
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Percentage of participants
  Improved Fibrosis Score | 24.8 | 42.3
  Stable Fibrosis Score | 52.9 | 39.8
  Worsened Fibrosis Score | 22.3 | 17.9

11. Secondary Outcome: Mean Change From Baseline in Activity and Fibrosis Scores Based on METAVIR Activity at Week 72
Description: METAVIR activity scores are categorised as histological activity (A) 0 = none; A1 = mild; A2 = moderate; A3 = severe where '0' being 'No activity' and '3' being 'the sever activity'. Changes in liver inflammation defined as Improved: Participants whose METAVIR activity score at up to Month-72 decreases by 1 or more units compared to baseline; stable: Participants whose METAVIR activity score at up to Month-72 is the same as the baseline score; worsened: Participants whose METAVIR activity score at up to Month-72 increases by 1 or more units compared to baseline. METAVIR fibrosis scores are categorised as fibrosis (F) 0 = no fibrosis; F1 = without septa; F 2 = with septa; F3 = many septa; F4 = cirrhosis where; '0' being the best and '4' being the worst. Decrease in score from baseline indicates improvement. The difference between study groups in change from baseline in activity and fibrosis scores based on METAVIR at week 72 was analysed.
Time Frame: From Baseline (Week 0) to Week 72
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Score on a scale
  Activity scores based on METAVIR | -0.34 (0.05) | -0.51 (0.05)
  Fibrosis scores based on METAVIR | 0.04 (0.07) | -0.12 (0.05)

12. Secondary Outcome: Percentage of Participants With Improved, Stable, and Worsened METAVIR Activity Score
Description: METAVIR activity scale included activity defines as, Improved: >= 1 category decrease in activity score; stable: no change in activity score; worsened: > = 1 category increase in activity score.
Time Frame: At Week 72
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Percentage of participants
  Stable Activity Score | 54.1 | 48.8
  Worsened Activity Score | 7.0 | 3.0
  Improved Activity Score | 38.9 | 48.3

13. Secondary Outcome: Percentage of Participants With Improved, Stable, and Worsened METAVIR Fibrosis Score
Description: METAVIR fibrosis score is categorized as, Improved: >= 1 category decrease in activity score; stable: no change in activity score; worsened: >= 1 category increase in activity score.
Time Frame: At Week 72
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Percentage of participants
  Stable Fibrosis Score | 71.3 | 66.2
  Worsened Fibrosis Score | 15.3 | 11.4
  Improved Fibrosis Score | 13.4 | 22.4

14. Secondary Outcome: Mean Change From Baseline in Fat Score at Week 72
Description: Grading categories for the fat scale were as follows: 1 = <5% hepatocytes; 2 = 6 - 33% hepatocytes; 3 = 34 - 66% hepatocytes; 4 = 67 - 100% hepatocytes.
Time Frame: From Baseline (Week 0) to Week 72
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Score on a scale | -0.15 (0.07) | -0.25 (0.06)

15. Secondary Outcome: Percentage of Participants With Improved, Stable and Worsened Fat Score From Baseline to Week 72
Description: Fat scores are categorised as Improved: > 1 category decrease in fat scale; stable: no change in fat scale; worsened: >= 1 category increase in fat scale.
Time Frame: From Baseline (Week 0) to Week 72
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Percentage of participants
  Stable Fat Score | 47.8 | 51.2
  Worsened Fat Score | 20.4 | 16.4
  Improved Fat Score | 31.8 | 32.3

16. Secondary Outcome: Percentage of Participants With Non-zero Nonalcoholic Steatohepatitis Score
Description: The Nonalcoholic Steatohepatitis (NASH) included an assessment of sinusoidal fibrosis, Mallory bodies, and hepatocyte ballooning (HB). Grading categories for the NASH scales were as: Sinusoidal fibrosis: 0 = absent; 1 = involvement of some lobules; 2 = involvement of most lobules, without diffuse interstitial sinusoidal collagen deposition; 3 = Involvement of most or all lobules;, with diffuse interstitial fibrosis involving some or most of the lobules Mallory bodies: 0 = absent; 1 = involvement of some lobules; 2 = involvement of most lobules; 3= involvement of most or all lobules; and Hepatocyte ballooning: 0 = absent; 1 = involvement of some lobules; 2 = involvement of most lobules; 3= involvement of most or all lobules.
Time Frame: At Week 72
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 157 | 201
Percentage of participants
  Sinusoidal Fibrosis Non-zero NASH Score at Week 72 | 19.1 | 18.4
  Mallory Bodies Non-zero NASH Score at Week 72 | 3.2 | 2.0
  HB Non-zero NASH Score at Week 72 | 19.7 | 9.5

17. Secondary Outcome: Mean Change in Fatigue Severity Scale Score and Fatigue Severity Scale Score Item 10 Visual Analog Scale Score From Baseline at Week 48 and Week 72
Description: The Fatigue Severity Scale (FSS) is a 10-item self-report questionnaire designed to assess tiredness, lack of energy, or total body give-out. Participants were to react to nine statements regarding fatigue over the previous 2 weeks, each on a scale (1 = completely agree, 7 = completely disagree). The FSS is the average of the scores on the 9 questions; ranging from 1-7, with lower scores indicating less fatigue. In addition, participants were to react to how much fatigue they had in the past 2 weeks by marking on a visual analogue scale (VAS) labelled at one end with "no fatigue" ('0' being the best) and at the other end with "greater fatigue" ('100' being the worst). Longer distance on the scale from "no fatigue" indicated "greater fatigue". FSS values are presented based on questionnaire and visual analog scale. FSS values at week 48 and 72 are presented based on questionnaire and visual analog scale.
Time Frame: Baseline (Week 0), Week 48 and Week 72
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 180 | 224
Score on a scale
  FSS Score,From Baseline At Week 48 (n=180,224) | 0.9 (0.15) | 1.5 (0.13)
  FSS Score,From Baseline At Week 72 (n=174,214) | -0.1 (0.15) | 0.1 (0.11)
  FSS VAS Score,From Baseline At Week 48 (n=177,221) | 14.8 (2.84) | 25.4 (2.09)
  FSS VAS Score,From Baseline At Week72 (n=173,212) | 1.9 (2.75) | -2.7 (1.57)
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; FSS Score of Latino VS Non-Latino White at week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; Study Group Difference = -0.65, 95% CI 2-sided [-0.96 to -0.33], Standard Error of Mean 0.162 — The estimated value is the difference of change from baseline in FSS scores at week 48 between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Latino vs Non-Latino White; FSS Score of Latino VS Non-Latino White at week 72; Test type: Superiority or Other; p = 0.0921, ANCOVA; Study Group Difference = -0.26, 95% CI 2-sided [-0.57 to 0.04], Standard Error of Mean 0.156 — The estimated value is the difference of change from baseline in FSS scores at week 72 between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 3: Comparison: Latino vs Non-Latino White; FSS VAS Score of Latino VS Non-Latino White at week 48; Test type: Superiority or Other; p = 0.0015, ANCOVA; Study Group Difference = -8.72, 95% CI 2-sided [-14.07 to -3.36], Standard Error of Mean 2.725 — The estimated value is the difference of change from baseline in FSS VAS scores at week 48 between Latino and Non-Latino White participants The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Latino vs Non-Latino White; FSS VAS Score of Latino VS Non-Latino White at week 72; Test type: Superiority or Other; p = 0.0421, ANCOVA; Study Group Difference = 4.83, 95% CI 2-sided [0.18 to 9.49], Standard Error of Mean 2.370 — The estimated value is the difference of change from baseline in FSS VAS scores at week 72 between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial

18. Secondary Outcome: Mean Change in 36-item Short Form Health Survey Total and Domain Scores From Baseline at Week 48 and 72
Description: The 36-item Short Form Health Survey (SF-36) is a 36-item self-report questionnaire that includes 8 domain scales The 8 domains are incorporated into 2 components: mental and physical. The mental component (MC) includes social functioning, role limitations-emotional, mental health, and vitality. The physical component (PC) includes physical functioning, role limitations-physical, bodily pain, and general health perception. Raw domain scores are transformed to a 0 to 100 scale, [0=worst score (or quality of life) and 100=best score]. Two summary scale scores were computed based on weighted combinations of the 8 domain scores (Physical and the Mental Component) where no minimum or maximum score; higher score indicate better health status. The difference between study groups in change from baseline in SF-36 score at week 48 and 72 was analysed.
Time Frame: Baseline (Week 0), Week 48 and Week 72
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 178 | 224
Score on a scale
  Standardized PC, At Week 48 (n=178,224) | -4.3 (0.75) | -8.4 (0.60)
  Standardized PC, At Week 72 (n=172,213) | -1.4 (0.71) | -1.8 (0.53)
  Standardized MC, At Week 48 (n=178,224) | -6.1 (0.77) | -6.3 (0.68)
  Standardized MC, At Week 72 (n=172,213) | -1.6 (0.73) | -0.7 (0.66)
Statistical Analysis 1: Comparison: Latino vs Non-Latino White; Standardized Physical Component of Latino VS Non-Latino White at week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; Study Group Difference = 3.49, 95% CI 2-sided [1.79 to 5.18], Standard Error of Mean 0.864 — The estimated value is the difference of change from baseline in standardized physical component score at week 48 between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 2: Comparison: Latino vs Non-Latino White; Standardized Physical Component of Latino VS Non-Latino White at week 72; Test type: Superiority or Other; p = 0.9047, ANCOVA; Study Group Difference = 0.10, 95% CI 2-sided [-1.49 to 1.68], Standard Error of Mean 0.808 — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Latino vs Non-Latino White; Standardized Mental Component of Latino VS Non-Latino White at week 48; Test type: Superiority or Other; p = 0.9286, ANCOVA; Study Group Difference = -0.08, 95% CI 2-sided [-1.88 to 1.71], Standard Error of Mean 0.914 — The estimated value is the difference of change from baseline in standardized mental component score at week 48 between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial
Statistical Analysis 4: Comparison: Latino vs Non-Latino White; Standardized Mental Component of Latino VS Non-Latino White at week 72; Test type: Superiority or Other; p = 0.1653, ANCOVA; Study Group Difference = -1.23, 95% CI 2-sided [-2.98 to 0.51], Standard Error of Mean 0.888 — The estimated value is the difference of change from baseline in standardized mental component score at week 72 between Latino and Non-Latino White participants. The 95% Confidence Interval is based on normal approximation to the binomial

19. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An adverse event could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing conditions that worsened during the study were reported as adverse events. A serious adverse event (SAE) was any untoward medical occurrence that at any dose results in death, is life threatening, requires hospitalization or prolongation of hospitalization, or results in disability/incapacity, or congenital anomaly/birth defect.
Time Frame: Up to Week 72
Population: The Safety Population included participants who received at least 1 dose of any study drug and had at least 1 post baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 299
Participants
  Any AEs | 264 | 292
  Any SAEs | 42 | 48

20. Secondary Outcome: Number of Participants With Marked Abnormal Laboratory Parameters
Description: The below table includes participants with marked abnormal lab parameters. Standard reference ranges include: Hematocrit: (fraction) 0.37 - 0.49, Hemoglobin 130 - 180 g/L, Platelets 150 - 350 10^9/L, White Blood Cell (WBC) 4.5 - 11.0 10^9/L, Lymphocytes 1.00 - 4.80 10^9/L, Neutrophils 1.80 - 7.70 10^9/L, Aspartate aminotransferase (AST) 0-40 U/L, ALT 0 - 55 U/L, Total bilirubin 0 - 17 μmol/L, Thyroxine T4 58 - 140 nmol/L, Thyroid Stimulating Hormone (TSH) 0.0 - 5.0 million units (mU)/L, Albumin 35.0 - 55.0 g/L, Chloride 100 - 108 mmol/L, Calcium 2.10 - 2.60 mmol/L, Phosphate 0.84 - 1.45 mmol/L, Uric acid 214 - 506 μmol/L.
Time Frame: Up to Week 72
Population: The Safety Population included participants who received at least 1 dose of any study drug and had at least 1 post baseline safety assessment. 'n'=number of evaluable participants available at specified time point.
Measure: Number; unit: Participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 299
Participants
  Hematocrit low (n=269,298) | 49 | 67
  Hemoglobin low (n=269,298) | 99 | 126
  Platelets, low (n=269,298) | 78 | 103
  WBC, high (n=269,298) | 2 | 7
  WBC low (n=269,298) | 192 | 253
  Lymphocytes low (n=269,298) | 80 | 159
  Neutrophils, high (n=269,298) | 7 | 15
  Neutrophils, low (n=269,298) | 208 | 261
  AST, high (n=269,296) | 51 | 47
  ALT, high (n=269,296) | 46 | 47
  Total bilirubin, high (n=269,296) | 4 | 6
  T4, high (n=17,16) | 2 | 2
  T4, low (n=17,16) | 8 | 4
  TSH, high (n=64,65) | 6 | 11
  Albumin, low (n=269,296) | 2 | 5
  Chloride, low (n=269,296) | 0 | 6
  Calcium, low (n=269,296) | 4 | 16
  Phosphate, high (n=269,296) | 16 | 18
  Phosphate, low (n=269,296) | 51 | 50
  Uric acid, high (n=269,296) | 12 | 9

21. Secondary Outcome: Number of Participants With Premature Withdrawals Due to Adverse Events or Laboratory Abnormalities
Description: The table below includes participants with premature withdrawals due to adverse events or laboratory abnormalities.
Time Frame: Up to Week 72
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Latino | Non-Latino White
Number analyzed (Participants) | 269 | 299
Participants
  Psychiatric disorders | 8 | 12
  General disorders | 4 | 5
  Blood and lymphatic system disorders | 3 | 6
  Gastrointestinal disorders | 2 | 4
  Nervous system disorders | 3 | 3
  Respiratory, thoracic and mediastinal disorders | 2 | 3
  Skin and subcutaneous tissue disorders | 1 | 3
  Eye disorders | 0 | 4
  Musculoskeletal and connective tissue disorders | 1 | 2
  Investigations | 3 | 0
  Infections and infestations | 1 | 1
  Injury, poisoning and procedural complications | 0 | 2
  Social circumstances | 0 | 2
  Cardiac disorders | 1 | 0
  Endocrine disorders | 1 | 0
  Vascular disorders | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An AE was therefore any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study drug.
Arm/Group | Latino | Non-Latino White
Serious Adverse Events (participants affected / at risk) | 42/269 | 48/299
Other Adverse Events (participants affected / at risk) | 256/269 | 290/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latino (N=269) | Non-Latino White (N=299)
Cellulitis (Infections and infestations) | 5 | 2
Pneumonia (Infections and infestations) | 0 | 4
Appendicitis (Infections and infestations) | 2 | 1
Abscess limb (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 4 | 4
Suicidal ideation (Psychiatric disorders) | 3 | 5
Suicide attempt (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 1
Bipolar II disorder (Psychiatric disorders) | 0 | 1
Homicidal ideation (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Cataract subcapsular (Eye disorders) | 0 | 1
Retinal exudates (Eye disorders) | 0 | 1
Retinal ischaemia (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous stasis (Vascular disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Haemobilia (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Activities of daily living impaired (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Latino (N=269) | Non-Latino White (N=299)
Fatigue (General disorders) | 167 | 205
PYREXIA (General disorders) | 67 | 86
INFLUENZA LIKE ILLNESS (General disorders) | 78 | 74
IRRITABILITY (General disorders) | 45 | 84
CHILLS (General disorders) | 50 | 57
PAIN (General disorders) | 40 | 43
INJECTION SITE REACTION (General disorders) | 18 | 25
INJECTION SITE ERYTHEMA (General disorders) | 8 | 23
ASTHENIA (General disorders) | 12 | 18
NAUSEA (Gastrointestinal disorders) | 84 | 117
DIARRHOEA (Gastrointestinal disorders) | 57 | 65
VOMITING (Gastrointestinal disorders) | 29 | 42
CONSTIPATION (Gastrointestinal disorders) | 22 | 22
ABDOMINAL PAIN (Gastrointestinal disorders) | 22 | 21
DYSPEPSIA (Gastrointestinal disorders) | 22 | 20
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 17 | 17
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 12 | 19
DRY MOUTH (Gastrointestinal disorders) | 11 | 20
STOMATITIS (Gastrointestinal disorders) | 7 | 23
INSOMNIA (Psychiatric disorders) | 91 | 140
DEPRESSION (Psychiatric disorders) | 69 | 79
ANXIETY (Psychiatric disorders) | 30 | 51
AGITATION (Psychiatric disorders) | 6 | 19
HEADACHE (Nervous system disorders) | 128 | 156
DIZZINESS (Nervous system disorders) | 46 | 59
DYSGEUSIA (Nervous system disorders) | 22 | 24
DISTURBANCE IN ATTENTION (Nervous system disorders) | 7 | 15
RASH (Skin and subcutaneous tissue disorders) | 62 | 97
ALOPECIA (Skin and subcutaneous tissue disorders) | 49 | 59
PRURITUS (Skin and subcutaneous tissue disorders) | 42 | 61
DRY SKIN (Skin and subcutaneous tissue disorders) | 34 | 51
MYALGIA (Musculoskeletal and connective tissue disorders) | 64 | 57
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 57 | 61
BACK PAIN (Musculoskeletal and connective tissue disorders) | 34 | 35
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 14 | 37
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 12 | 19
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 18 | 12
COUGH (Respiratory, thoracic and mediastinal disorders) | 43 | 74
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 24 | 57
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 22 | 16
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 | 27
ANAEMIA (Blood and lymphatic system disorders) | 59 | 73
NEUTROPENIA (Blood and lymphatic system disorders) | 31 | 40
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 24 | 20
NASOPHARYNGITIS (Infections and infestations) | 15 | 20
SINUSITIS (Infections and infestations) | 7 | 20
BRONCHITIS (Infections and infestations) | 7 | 18
INFLUENZA (Infections and infestations) | 6 | 16
DECREASED APPETITE (Metabolism and nutrition disorders) | 27 | 48
ANOREXIA (Metabolism and nutrition disorders) | 35 | 20
WEIGHT DECREASED (Investigations) | 32 | 49
VISION BLURRED (Eye disorders) | 16 | 29
DRY EYE (Eye disorders) | 4 | 15
HYPERTENSION (Vascular disorders) | 8 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.